CLINICAL TRIAL: NCT00896896
Title: Immunoreactivity to Cetuximab in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC HN 0668; VU-VICC-HN-0668
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Colorectal Cancer; Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage I adenoid cystic carcinoma of the oral cavity; stage I basal cell carcinoma of the lip; stage I mucoepidermoid carcinoma of the oral cavity; stage I squamous cell carcinoma of the lip and oral cavity; stage I verrucous carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage II basal cell carcinoma of the lip; stage II mucoepidermoid carcinoma of the oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage II verrucous carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III basal cell carcinoma of the lip; stage III mucoepidermoid carcinoma of the oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV basal cell carcinoma of the lip; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV verrucous carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; recurrent basal cell carcinoma of the lip; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; stage I lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent salivary gland cancer; recurrent squamous cell carcinoma of the oropharynx; recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Immunologic Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: immunologic technique — Sera from head and neck cancer or colorectal cancer patients who were treated with cetuximab will be obtained from Tumor Tissue Repository
  Other Names: None indicated
Other: laboratory biomarker analysis — Sera from head and neck cancer or colorectal cancer patients who were treated with cetuximab will be obtained from Tumor Tissue Repository
  Other Names: None indicated

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory may help doctors predict which patients will develop hypersensitivity to cetuximab.

PURPOSE: This research study is looking at hypersensitivity to cetuximab in patients with head and neck cancer or advanced colorectal cancer previously treated with cetuximab.

DETAILED DESCRIPTION:
OBJECTIVES:

* To examine serum samples from patients with head and neck cancer or advanced colorectal cancer previously treated with cetuximab for the presence of antibodies against cetuximab.

OUTLINE: Serum samples are examined by immunoreactivity screening of IgE, IgG, IgA, and IgM antibodies and complement reaction.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following:

  * Head and neck cancer
  * Advanced colorectal cancer
* Previously treated with cetuximab
* Serum samples available from patients enrolled in one of the following clinical trials:

  * VU-VICC-GI-0410 (colorectal cancer)
  * VU-VICC-GI-0622 (colorectal cancer)
  * VU-VICC-HN-0356 (head and neck cancer)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head and neck cancer or colorectal cancer patients who were treated with cetuximab
Sampling Method: Non-Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Identification of antibodies (e.g., IgE, IgG, IgA, and IgM) against cetuximab | Until all samples are collected.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Murphy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center